CLINICAL TRIAL: NCT01268683
Title: A Multi-Center, Prospective, Open Label, Phase IIa Trial of RP-1127 (Glyburide for Injection) in Patients With a Severe Anterior Circulation Ischemic Stroke Who Are Likely to Experience Clinically Significant Brain Swelling.
Brief Title: Glyburide Advantage in Malignant Edema and Stroke Pilot
Acronym: GAMES-PILOT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Remedy Pharmaceuticals, Inc. (Industry)
Collaborators: University of Maryland (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RPI 201
Record Dates: First submitted 2010-12-29; First posted 2010-12-31 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Glyburide; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Glyburide for Injection (Experimental): This arm is administered a glyburide bolus followed by continuous infusion of glyburide for 72 hours
  Interventions: Drug: Glyburide for Injection

INTERVENTIONS:
Drug: Glyburide for Injection — Administered as specified in the treatment arm.
  Other Names: RP-1127; glibenclamide; glybenclamide

SUMMARY:
The primary objective of this study is to assess the feasibility of enrolling, evaluating, and treating with glyburide for injection severe anterior circulation ischemic stroke participants, whether or not treated with standard of care intravenous (IV) recombinant tissue plasminogen activator (rtPA). Participants must be between 18-80 years of age, must have a baseline diffusion weighted image (DWI) lesion volume 82 -210 centimeters cubed (cm3), and time from symptom onset to start of study infusion must be ≤10 hour(hr). The secondary objectives are to assess the initial safety and tolerability, and pharmacokinetics (PK) /pharmacodynamics (PD) of glyburide in severe stroke participants, as well as to compare the clinical and magnetic resonance imaging (MRI) outcome data to benchmark data derived from published literature.

DETAILED DESCRIPTION:
This is a multi-center, prospective, open label, phase IIa trial of glyburide for injection in 10 participants with a severe anterior circulation ischemic stroke who are likely to experience clinically significant brain swelling.

Participants will receive glyburide, delivered as an IV bolus followed by an IV infusion for 72 hours.

Participants will have a baseline (pretreatment) MRI scan as standard of care, and three follow up MRI scans (at 24+12 hours, 48+12 hours, and 72±12 hours). Since recanalization may have an effect on outcome, the results of vascular studies, obtained as part of standard of care and defined as CTA, MRA or catheter angiography of the head and neck, will be recorded. Additionally, clinical endpoints such as the National Institutes of Health Stroke Scale (NIHSS), Glasgow Coma Scale (GCS) and Full Outline of UnResponsiveness Score (FOUR) Score (baseline, 24±12 hour, 48±12 hour, 72±12 hour and 7±1 days) and Modified Rankin Scale (mRS) (30±5 days and 90±7 days) will be assessed. Safety parameters will be assessed through Day 7 or discharge (whichever is sooner), and then again at Day 30±5 and Day 90±7.

Study participation is expected to last 90±7 days.

ELIGIBILITY:
Key Inclusion Criteria:

* A clinical diagnosis of acute ischemic stroke in the MCA or MCA/ACA territory.
* Pre-morbid mRS 0 - 1.
* A baseline DWI lesion between 82 cm3 and 210 cm3 on MRI.
* Patients treated with IV rtPA should meet established criteria for IV rtPA administration in the 0-3 and 3-4.5 hr time periods, respectively.
* The time to the start of infusion of study compound must be ≤ 10 hr after time of symptom onset
* Age ≥18 years and ≤70 years.
* Provision of written informed consent by the patient or from a legally authorized representative according to institutional guidelines and national regulations.

Key Exclusion Criteria:

* Evidence from imaging or pre-enrollment investigation of any diagnosis other than acute ischemic stroke likely to cause the presenting symptoms and signs.
* Commitment to decompressive craniectomy (DC) prior to enrollment, or follow-ing enrollment and prior to start of study compound.
* Treatment with IA rtPA or by mechanical means for clot disruption or with hypo-thermia.
* Patients unable to tolerate MRI scanning, e.g. those with pacemakers or automatic defibrillators.
* Pre-morbid mRS ≥ 2.
* Clinical signs of herniation, e.g. one or two dilated, fixed pupils; unconsciousness (i.e., ≥ 2 on item 1a on the NIHSS); loss of other brain stem reflexes attributable to herniation according to the investigator's judgment.
* CT or MRI evidence of hemorrhage or anteroseptal/pineal shift greater ≥2 mm prior to enrollment.
* Rapidly improving symptoms.
* Severe renal disorder from the patient's history (e.g. dialysis) or eGFR of < 30 mL/min/1.73 m2.
* Severe liver disease or ALT, AST, or bilirubin >2 times normal.
* Blood glucose <55 mg/dL at enrollment or immediately prior to administration of RP-1127, or a clinically significant history of hypoglycemia.
* Diagnosis of decompensated heart failure (e.g. clinical diagnosis of pulmonary edema, chest x-ray consistent with heart failure, tachypnea > 20, etc.)
* Sulfonylurea treatment within 30 days.
* Known allergy to sulfa or specific allergy to sulfonylurea drugs.
* Known G6PD enzyme deficiency.
* Pregnancy or breast-feeding. Women must be either post-menopausal (judged by the investigator), permanently sterilized or, if of childbearing age, must have a negative test for pregnancy obtained before enrollment.
* Patients already enrolled in a non-observation-only stroke study, or with life-expectancy <3 months not related to current stroke, or those unlikely to be com-pliant with follow up.
* Patients who, in the opinion of the investigator, are not suitable for the study (reason to be documented).

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-05-26 (Actual); Primary Completion 2012-06-07 (Actual); Study Completion 2012-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Remedy Pharmaceuticals
Locations (4):
- United States (4):
  - Rush University Medical Center, Chicago, Illinois
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Kimberly WT, Battey TW, Pham L, Wu O, Yoo AJ, Furie KL, Singhal AB, Elm JJ, Stern BJ, Sheth KN. Glyburide is associated with attenuated vasogenic edema in stroke patients. Neurocrit Care. 2014 Apr;20(2):193-201. doi: 10.1007/s12028-013-9917-z. PMID 24072459
- [Background] Sheth KN, Kimberly WT, Elm JJ, Kent TA, Yoo AJ, Thomalla G, Campbell B, Donnan GA, Davis SM, Albers GW, Jacobson S, del Zoppo G, Simard JM, Stern BJ, Mandava P. Exploratory analysis of glyburide as a novel therapy for preventing brain swelling. Neurocrit Care. 2014 Aug;21(1):43-51. doi: 10.1007/s12028-014-9970-2. PMID 24671831
- [Result] Sheth KN, Kimberly WT, Elm JJ, Kent TA, Mandava P, Yoo AJ, Thomalla G, Campbell B, Donnan GA, Davis SM, Albers GW, Jacobson S, Simard JM, Stern BJ. Pilot study of intravenous glyburide in patients with a large ischemic stroke. Stroke. 2014 Jan;45(1):281-3. doi: 10.1161/STROKEAHA.113.003352. Epub 2013 Nov 5. PMID 24193798

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 2011, and May 2012, ten subjects were enrolled and treated at University of Maryland and the Massachusetts General Hospital within 9.6 months at 2 sites.
Groups:
- RP-1127 (Glyburide for Injection): RP-1127 (Glyburide for injection) : Bolus plus 72 hour IV infusion
Period: Overall Study
Arm/Group | RP-1127 (Glyburide for Injection)
Started | 10
Completed | 8
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | RP-1127 (Glyburide for Injection)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 50.5 [25 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Rate of Enrollment
Description: The number of months to enroll 10 participants.
Time Frame: Day 1
Measure: Number; unit: Months
Arm/Group | RP-1127 (Glyburide for Injection)
Number analyzed (Participants) | 10
Months | 9.6

2. Primary Outcome: Percentage of Enrolled Participants to Screened Participants
Time Frame: Day 1
Measure: Number; unit: Percentage of Participants
Arm/Group | RP-1127 (Glyburide for Injection)
Number analyzed (Participants) | 175
Percentage of Participants | 5.7

3. Primary Outcome: Percentage of Participants Completing 90-Day Follow-Up
Time Frame: Day 90
Measure: Number; unit: Percentage of Participants
Arm/Group | RP-1127 (Glyburide for Injection)
Number analyzed (Participants) | 10
Percentage of Participants | 80

4. Primary Outcome: Percentage of Dose Reductions/ Dose Suspensions
Time Frame: Up to Day 3
Measure: Number; unit: Percentage of Participants
Arm/Group | RP-1127 (Glyburide for Injection)
Number analyzed (Participants) | 10
Percentage of Participants | 0

5. Primary Outcome: Percentage of Participants With All Four MRI Assessments Per Protocol
Time Frame: Up to Day 3
Measure: Number; unit: Percentage of Participants
Arm/Group | RP-1127 (Glyburide for Injection)
Number analyzed (Participants) | 10
Percentage of Participants | 90

6. Primary Outcome: Number of MRI Assessments Per Participant
Time Frame: Up to Day 3
Measure: Mean (Full Range); unit: Number of MRIs
Arm/Group | RP-1127 (Glyburide for Injection)
Number analyzed (Participants) | 10
Number of MRIs | 3.9 [3 to 4]

7. Primary Outcome: Percentage of Participants Requiring One or More Hypoglycemia Treatments
Time Frame: Up to Day 4
Measure: Number; unit: Percentage of Participants
Arm/Group | RP-1127 (Glyburide for Injection)
Number analyzed (Participants) | 10
Percentage of Participants | 0

8. Primary Outcome: Percentage of Participants With Pre-specified Adverse Events Associated With Glyburide According to Protocol
Time Frame: Up to Day 4
Measure: Number; unit: Percentage of Participants
Arm/Group | RP-1127 (Glyburide for Injection)
Number analyzed (Participants) | 10
Percentage of Participants | 0

9. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: Adverse Events (AE's) of special interest (cardiac events, difficulty controlling blood sugar, liver problems, and blood disorders, including anemia) will be followed for 30 days and all Severe Adverse Events (SAE's) will be followed for 90 days. SAE's and AE's were reviewed, and the number of participants with unanticipated adverse events, or drug-related SAE's were assessed.
Time Frame: Up to Day 90
Measure: Number; unit: Number of Participants
Arm/Group | RP-1127 (Glyburide for Injection)
Number analyzed (Participants) | 10
Number of Participants
  Adverse Events | 10
  Serious Adverse Events | 3

10. Secondary Outcome: Infarcted Hemisphere Volume
Time Frame: Baseline, Day 1, Day 2, and Day 3
Population: The number analyzed varies due to only MRIs of good quality being analyzed.
Measure: Mean (Standard Deviation); unit: Centimeters cubed (cm^3)
Arm/Group | RP-1127 (Glyburide for Injection)
Number analyzed (Participants) | 10
Centimeters cubed (cm^3)
  Baseline | 135.20 (27.19)
  Day 1: number analyzed (Participants) | 9
  Day 1 | 156.78 (35.09)
  Day 2: number analyzed (Participants) | 8
  Day 2 | 165.38 (34.17)
  Day 3: number analyzed (Participants) | 7
  Day 3 | 181.71 (33.90)

11. Secondary Outcome: Absolute Diffusion Weighted Imaging (DWI) Lesion Volume
Time Frame: Baseline, Day 1, Day 2, and Day 3
Population: The number analyzed varies due to only MRIs of good quality being analyzed.
Measure: Mean (Standard Deviation); unit: Cm^3
Arm/Group | RP-1127 (Glyburide for Injection)
Number analyzed (Participants) | 10
Cm^3
  Baseline: number analyzed (Participants) | 9
  Baseline | 101.76 (22.57)
  Day 1: number analyzed (Participants) | 9
  Day 1 | 141.62 (44.05)
  Day 2: number analyzed (Participants) | 8
  Day 2 | 152.31 (49.26)
  Day 3: number analyzed (Participants) | 6
  Day 3 | 169.73 (54.28)

12. Secondary Outcome: Change From Baseline in DWI Lesion Volume
Time Frame: Baseline, Day 1, Day 2, and Day 3 (Day 3 reported)
Measure: Mean (Standard Deviation); unit: Cm^3
Arm/Group | RP-1127 (Glyburide for Injection)
Number analyzed (Participants) | 10
Cm^3 | 60.30 (41.37)

13. Secondary Outcome: Midline Shift
Time Frame: Baseline, Day 1, Day 2, and Day 3
Population: The number analyzed varies due to only MRIs of good quality being analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | RP-1127 (Glyburide for Injection)
Number analyzed (Participants) | 10
Millimeters (mm)
  Baseline: number analyzed (Participants) | 9
  Baseline | 0.56 (1.13)
  Day 1: number analyzed (Participants) | 9
  Day 1 | 2.00 (2.29)
  Day 2: number analyzed (Participants) | 8
  Day 2 | 2.63 (1.41)
  Day 3: number analyzed (Participants) | 6
  Day 3 | 2.50 (2.17)

14. Secondary Outcome: Ipsilateral Ventricle Volume
Time Frame: Baseline, Day 1, Day 2, and Day 3
Population: The number analyzed varies due to only MRIs of good quality being analyzed.
Measure: Mean (Standard Deviation); unit: Cm^3
Arm/Group | RP-1127 (Glyburide for Injection)
Number analyzed (Participants) | 10
Cm^3
  Baseline: number analyzed (Participants) | 9
  Baseline | 11.78 (5.98)
  Day 1: number analyzed (Participants) | 9
  Day 1 | 9.25 (4.74)
  Day 2: number analyzed (Participants) | 8
  Day 2 | 8.92 (4.30)
  Day 3: number analyzed (Participants) | 6
  Day 3 | 10.07 (6.38)

15. Secondary Outcome: Frequency of Hemorrhagic Events
Time Frame: Day 1, Day 2, and Day 3
Measure: Number; unit: Number of Events
Arm/Group | RP-1127 (Glyburide for Injection)
Number analyzed (Participants) | 10
Number of Events
  Hemorrhagic Infarction Type 1 | 3
  Hemorrhagic Infarction Type 2 | 8
  Parenchymal Hematoma Type 1 | 0
  Parenchymal Hematoma Type 2 | 0

16. Secondary Outcome: National Institute of Health Stroke Scale (NIHSS) Score
Description: The NIHSS is composed of 11 categories, each of which is scored between 0 and 4. A score of 0 indicates normal function, a higher score indicates more impairment. Category scores are summed to generate the total NIHSS score (possibles scores range from 0-42).
Time Frame: Baseline, Day 1, Day 2, Day 3, and Day 7
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | RP-1127 (Glyburide for Injection)
Number analyzed (Participants) | 10
Score on a Scale
  Baseline | 17.8 (5.92)
  Day 1 | 18.4 (8.47)
  Day 2 | 15.6 (5.42)
  Day 3 | 16.2 (5.35)
  Day 7 | 13.9 (5.51)

17. Secondary Outcome: Glasgow Coma Scale (GCS) Score
Description: The GCS is scored on a scale between 3 and 15 (3 = the worst, and 15 = best). It is composed of three parameters : Best Eye Response (scored on a scale of 1-4), Best Verbal Response (scored on a scale of 1-5), Best Motor Response (scored on a scale of 1-6)
Time Frame: Baseline, Day 1, Day 2, Day 3, and Day 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | RP-1127 (Glyburide for Injection)
Number analyzed (Participants) | 10
Score on a scale
  Baseline | 12.5 (2.51)
  Day 1 | 11.9 (2.64)
  Day 2 | 12.5 (1.96)
  Day 3 | 12.8 (2.20)
  Day 7 | 13.5 (1.58)

18. Secondary Outcome: Full Outline of UnResponsiveness (FOUR) Score
Description: The FOUR Score is a 17-point scale (with potential scores ranging from 0 - 16). Decreasing FOUR Score is associated with worsening level of consciousness. The FOUR Score assesses four domains of neurological function: eye responses, motor responses, brainstem reflexes, and breathing pattern.
Time Frame: Baseline, Day 1, Day 2, Day 3, and Day 7
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | RP-1127 (Glyburide for Injection)
Number analyzed (Participants) | 10
Score on a Scale
  Baseline | 15.1 (1.10)
  Day 1 | 14.5 (2.32)
  Day 2 | 14.6 (2.27)
  Day 3 | 14.6 (1.65)
  Day 7 | 14.8 (1.99)

19. Secondary Outcome: Number of Participants Requiring Decompressive Craniectomy (DC)
Time Frame: Up to Day 90
Measure: Number; unit: Number of Participants
Arm/Group | RP-1127 (Glyburide for Injection)
Number analyzed (Participants) | 10
Number of Participants | 2

20. Secondary Outcome: Number of Participants With a Modified Rankin Scale (mRS) Score ≤ 4
Description: The mRS scale runs from 0-6, the scoring is as follows: 0 - No symptoms, 1 - No significant disability, 2 - Slight disability, 3 - Moderate disability, 4 - Moderately severe disability, 5 - Severe disability, 6 - Dead
Time Frame: Day 30, Day 90
Population: The number analyzed varies due to participants not completing follow up.
Measure: Number; unit: Number of Participants
Arm/Group | RP-1127 (Glyburide for Injection)
Number analyzed (Participants) | 10
Number of Participants
  Day 30 | 9
  Day 90: number analyzed (Participants) | 9
  Day 90 | 8

ADVERSE EVENTS:
Time Frame: Up to 90 Days
Arm/Group | RP-1127 (Glyburide for Injection)
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RP-1127 (Glyburide for Injection) (N=10)
Brain herniation (Nervous system disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RP-1127 (Glyburide for Injection) (N=10)
Agitation (Nervous system disorders) | 3
Alcohol withdrawal syndrome (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Staphylococcal bacteraemia (Infections and infestations) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Depression (Psychiatric disorders) | 1
Blood glucose decreased (Investigations) | 1
Dry eyes (Eye disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Endocrine disorders) | 1
Hypertension (Vascular disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Insomnia (Nervous system disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Pyrexia (General disorders) | 1
Transaminase increased (Investigations) | 1
Urinary tract infection (Infections and infestations) | 4
Hypovitaminosis (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 2
Agitation (Psychiatric disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Vision blurred (Nervous system disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 1
Open wound (Injury, poisoning and procedural complications) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 8
Pain (General disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 1
Central pain syndrome (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 1
Brain herniation (Nervous system disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The trial was a single arm; there is thus no placebo to compare RP-1127 to.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No